CLINICAL TRIAL: NCT05489094
Title: The Impact of Nutrition Education and Milk Provision in Fueling the Progress of 1 - 3 Years Old Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Danone Specialized Nutrition Indonesia (Industry)
Collaborators: Indonesian Nutrition Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 270422
Record Dates: First submitted 2022-07-26; First posted 2022-08-05 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized non blinded and controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): First group will be given nutrition education and iron intake from growing up milk approximately 2 - 3 servings/day for four months intervention period
  Interventions: Combination Product: Nutrition Education and Growing Up Milk for 1 - 3 years old
- Control Group (Placebo Comparator): Second group will be given nutrition education only for four months intervention period
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Combination Product: Nutrition Education and Growing Up Milk for 1 - 3 years old — Nutrition education is a basic information related balanced nutrition for 1 - 3 children including the details of food types and calories. while Intervention product is formulated to deliver macro- and micronutrients as part of the dietary intake for children at 1-3 years old with Iron-C formula
  Arms: Intervention Group
Behavioral: Nutrition Education — Nutrition education is a basic information related balanced nutrition for 1 - 3 children including the details of food types and calories.
  Arms: Control Group

SUMMARY:
The study will be conducted by the Indonesia Nutrition Association that led by a Principle Investigator and supported by the study team consisted of Nutritionists.

The aims of the study are to reduce iron deficiency by increasing iron intake in children 1-3 years by providing interventions in the form of increasing iron intake from growing up milk for four months and nutrition education for the intervention group and nutrition education only for the control group.

DETAILED DESCRIPTION:
The study will be conducted by the Indonesia Nutrition Association that led by a Principle Investigator and supported by the study team consisted of Nutritionists.

The aim of the study is to reduce iron deficiency by increasing iron intake in children 1-3 years (min 40%) by providing interventions in the form of increasing iron intake from growing up milk and nutrition education for the intervention group and nutrition education only for the control group for four months intervention period.

The subject for the study is 2 x 98 children for a cluster randomization control trial study residing in Kampung Melayu, East Jakarta. After signed informed consent had been obtained from parents/caretakers, baseline characteristics (demographics, medical history, pre-existing conditions, weight, and height) were collected and recorded. Children that have passed the requirements to be included and not to be excluded based on inclusion and exclusion criteria will be collected and recorded their data based on the protocol.

All children in the intervention group will be receiving nutrition education and growing up milk approximately 2-3 servings/day during the intervention period, whereas those who are in the control group will receive only nutrition education. Their data will be collected and recorded for the study.

During the intervention period, in a regular period, children in the study, will be measured on parameters that are stated above. Screening, enrolment, baseline measurements, subsequent assessments at 1, 2, 3, and 4 months of intervention will be done at the community health center in Jakarta. The monitoring to ensure adherent to the intervention will be conducted via home visits by health workers.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy Indonesian children
* Age 12 - 32 months at baseline visit
* Willing to take min 2 serving of study product per day
* Daily Iron intake less than 80% of Indonesian RDA (<5.6 mg/day)
* Planning to reside in the study area during the next 4 months
* Written informed consent by parent(s) or legally acceptable representative (in ICF there is statement that both are agree that child participate in the study)

Exclusion Criteria:

* Having Hb <8 g/dL using Hemocue
* Having cow's milk allergy, galactosemia, conditions needing a special diet, like major renal and hepatic dysfunction, major gastrointestinal intolerance (e.g., severe vomiting, severe diarrhea), investigator's uncertainty about the willingness or ability of the child/carer to comply with the protocol requirements, participation in any other study within two weeks prior to entry into the study

Ages: 12 Months to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Impact of milk provision on change from baseline of daily iron intake at 4 month in intervention group vs control group | at baseline and at 4 months after baseline (visit4)
  To know the impact of milk provision on change of daily iron intake using 24h recall and semi quantitative food frequency questionnaire in intervention group vs control group

SECONDARY OUTCOMES:
Impact of milk provision on the adequacy of iron intake based on percentage of recommended daily allowance | baseline
  To know the adequacy of iron intake based on percentage of recommended daily allowance at baseline in intervention group vs control group
Impact of milk provision on the adequacy of iron intake based on percentage of recommended daily allowance | 1 month after baseline (visit1)
  To know the adequacy of iron intake based on percentage of recommended daily allowance at 1 month in intervention group vs control group
Impact of milk provision on the adequacy of iron intake based on percentage of recommended daily allowance | 2 months after baseline (visit2)
  To know the adequacy of iron intake based on percentage of recommended daily allowance at 2 months in intervention group vs control group
Impact of milk provision on the adequacy of iron intake based on percentage of recommended daily allowance | 3 months after baseline (visit3)
  To know the adequacy of iron intake based on percentage of recommended daily allowance at 3 months in intervention group vs control group
Impact of milk provision on the adequacy of iron intake based on percentage of recommended daily allowance | 4 months after baseline (visit4)
  To know the adequacy of iron intake based on percentage of recommended daily allowance at 4 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Energy in kcal) | baseline
  To know the average daily nutrients intake (Energy in kcal) at baseline in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) | baseline
  To know the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) at baseline in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) | baseline
  To know the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) at baseline in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) | baseline
  To know the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) at baseline in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Energy in kcal) | 1 month after baseline (visit1)
  To know the average daily nutrients intake (Energy in kcal) at 1 month in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) | 1 month after baseline (visit1)
  To know the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) at 1 month in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) | 1 month after baseline (visit1)
  To know the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) at 1 month in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) | 1 month after baseline (visit1)
  To know the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) at 1 month in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Energy in kcal) | 2 months after baseline (visit2)
  To know the average daily nutrients intake (Energy in kcal) at 2 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) | 2 months after baseline (visit2)
  To know the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) at 2 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) | 2 months after baseline (visit2)
  To know the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) at 2 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) | 2 months after baseline (visit2)
  To know the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) at 2 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Energy in kcal) | 3 months after baseline (visit3)
  To know the average daily nutrients intake (Energy in kcal) at 3 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) | 3 months after baseline (visit3)
  To know the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) at 3 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) | 3 months after baseline (visit3)
  To know the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) at 3 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) | 3 months after baseline (visit3)
  To know the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) at 3 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Energy in kcal) | 4 months after baseline (visit4)
  To know the average daily nutrients intake (Energy in kcal) at 4 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) | 4 months after baseline (visit4)
  To know the average daily nutrients intake (Protein, Carbohydrate, Fat, Fiber & DHA in g) at 4 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) | 4 months after baseline (visit4)
  To know the average daily nutrients intake (Fe, Ca, P, Zn, Mg, Vit B6 & Vit E in mg) at 4 months in intervention group vs control group
Impact of milk provision on the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) | 4 months after baseline (visit4)
  To know the average daily nutrients intake (Folic Acid, Vit A, Vit C, Vit D & Vit B12 in μg) at 4 months in intervention group vs control group
Impact of milk provision on Total hemoglobin Level (SpHb) level using Masimo device | baseline
  To know the hemoglobin level at baseline in intervention group vs control group
Impact of milk provision on Total hemoglobin Level (SpHb) level using Masimo device | 4 months after baseline (visit4)
  To know the hemoglobin level at 4 months in intervention group vs control group
Impact of milk provision on nutritional status (weight, height - WAZ, HAZ, and WHZ) | baseline
  To know the nutritional status (weight, height - WAZ, HAZ, and WHZ) at baseline in intervention group vs control group
Impact of milk provision on nutritional status (weight, height - WAZ, HAZ, and WHZ) | 1 month after baseline (visit1)
  To know the nutritional status (weight, height - WAZ, HAZ, and WHZ) at 1 month in intervention group vs control group
Impact of milk provision on nutritional status (weight, height - WAZ, HAZ, and WHZ) | 2 months after baseline (visit1)
  To know the nutritional status (weight, height - WAZ, HAZ, and WHZ) at 2 months in intervention group vs control group
Impact of milk provision on nutritional status (weight, height - WAZ, HAZ, and WHZ) | 3 months after baseline (visit1)
  To know the nutritional status (weight, height - WAZ, HAZ, and WHZ) at 3 months in intervention group vs control group
Impact of milk provision on nutritional status (weight, height - WAZ, HAZ, and WHZ) | 4 months after baseline (visit1)
  To know the nutritional status (weight, height - WAZ, HAZ, and WHZ) at 4 months in intervention group vs control group

CONTACTS AND LOCATIONS:
Overall Officials: Dr. dr. Dian N Chandra, M.Gizi, Principal Investigator — Indonesian Nutrition Association (INA)

IPD SHARING:
Plan to Share IPD: No